CLINICAL TRIAL: NCT01624831
Title: Social Cognition in Longstanding Psychosis
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Nicholas Breitborde, Assistant Professor, Department of Psychiatry, University of Arizona
Other Study IDs: U. Az IRB 11-0567-02
Record Dates: First submitted 2011-11-07; First posted 2012-06-21 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder With Psychotic Features; Major Depression With Psychotic Features; Psychosis Not Otherwise Specified (NOS)
Keywords: Psychosis; schizophrenia; schizoaffective disorder; Bipolar disorder with psychotic features; Major depression with psychotic features; Psychosis NOS; Social Cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals with Longstanding Psychosis: Individuals with symptoms of psychosis that have been present for 5 or more years

SUMMARY:
In the current study, the investigators propose to measure the five domains of social cognition identified by the National Institute of Mental Health (NIMH) as relevant to individuals with psychosis (i.e., theory of mind, attribution style, emotion recognition, social perception, and social knowledge). The investigators will also explore the association between different domains of social cognition and outcomes relevant to psychotic disorder (e.g., symptomatology, social functioning, and vocational functioning).

DETAILED DESCRIPTION:
There is growing evidence that individuals with longstanding psychotic disorders suffer from deficits in social cognition (i.e., the cognitive skills needed to successfully navigate social interactions). However, to date, there have been few attempts to measure multiple components of social cognition within the same population of individuals with psychosis. Thus, the interrelationships between various aspects of social cognition remain unclear. In the current study, the investigators propose to measure the five domains of social cognition identified by NIMH as relevant to individuals with psychosis (i.e., theory of mind, attribution style, emotion recognition, social perception, and social knowledge). The investigators will also explore the association between different domains of social cognition and outcomes relevant to psychotic disorder (e.g., symptomatology, social functioning, and vocational functioning).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a schizophrenia spectrum disorder or an affective disorder with psychotic features per the Diagnostic and Statistical Manual of Mental Disorders-IV-Text Revised (DSM-IV-TR) criteria using the Structured Clinical Interview for the DSM-IV.
* Duration of psychotic symptoms greater than or equal to 5 years determined using the Symptom Onset in Schizophrenia Inventory
* Age 18-75
* No evidence of mental retardation.
* Able to provide informed consent as evidenced by passing the informed consent quiz with a score of 80% or greater.
* Fluent in English as assessed per self-report from participant

Exclusion Criteria:

* Unwilling or unable to complete study assessments (e.g., unable to read self-report questionnaires)
* Subject is currently pregnant per subject's report

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with longstanding psychotic disorder (i.e., 5 years or longer in duration)
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Emotion Recognition | Baseline and 6 months
  Change from baseline to 6 month assessment in ability to recognize emotions displayed by others assessed using the Facial Emotion Identification Test
Attribution Style | Baseline and 6 months
  Change from baseline to 6 month assessment in tendency to attribute events that occur to situational, personal, or internal factors assessed using the Internal, Personal, and Situational Attributions Questionnaire
Social Perception | Baseline and 6 months
  Change from baseline to 6 month assessment in ability to understand concrete and abstract components of everyday social interactions assessed using the Social Cues Recognition Test
Social Knowledge | Baseline and 6 months
  Change from baseline to 6 month assessment in knowledge of goals and actions associated with familiar and unfamiliar social activities assessed using the Situational Features Recognition Test
Theory of Mind | Baseline and 6 months
  Change from baseline to 6 month assessment in ability to identify the mental states of other individuals assessed using the Hinting Test

SECONDARY OUTCOMES:
Anxiety | Baseline and 6 months
  Change from baseline to 6 month assessment in anxiety assessed using the Beck Anxiety Inventory
Depression | Baseline and 6 months
  Change from baseline to 6 month assessment in depression assessed using the Beck Depression Inventory
Psychosis | Baseline and 6 months
  Change from baseline to 6 month assessment in severity of positive and negative psychotic symptoms assessed using the Positive and Negative Syndrome Scale
Social Functioning | Baseline and 6 months
  Change from baseline to 6 month assessment in level of social functioning assessed using the Social Functioning Scale
Service Utilization | Baseline and 6 months
  Change from baseline to 6 month assessment in utilization of medical services assessed using the Service Utilization Record Form
Self-Determination Needs Satisfaction | Baseline and 6 months
  Change from baseline to 6 month assessment in ability to fulfill basic needs for autonomy, competence, and relatedness assessed using the Basic Psychological Needs Scale
Locus of Control | Baseline and 6 months
  Change from baseline to 6 month assessment in perception of one's ability to control events in the environment assessed using the Multidimensional Locus of Control Scale
Cognitive representation of illness | Baseline and 6 months
  Change from baseline to 6 month assessment in understanding of nature of psychotic illness assessed using the Illness Perception Questionnaire
Emotional Awareness | Baseline and 6 months
  Change from baseline to 6 month assessment in awareness of one's own emotions as well as emotions of others assessed using the Levels of Emotional Awareness Scale
Mindfulness | Baseline and 6 months
  Change from baseline to 6 month assessment in awareness and acceptance of feelings and events assessed using the Philadelphia Mindfulness Scale
Medication adherence | Baseline and 6 months
  Change from baseline to 6 month assessment in adherence to psychiatric medication assessed using the Medication Adherence Rating Scale
Neuropsychological functioning | Baseline and 6 months
  Change from baseline to 6 month assessment in neuropsychological functioning assessed using the MATRICS Consensus Cognitive Battery
Social Support | Baseline and 6 months
  Change from baseline to 6 month assessment in level of social support assessed using the Measure of Perceived Support
Illness Uncertainty | Baseline and 6 months
  Change from baseline to 6 month assessment in uncertainty with regard to cause, course, and treatment of illness assessed using the Mischel Uncertainty in Illness Scale
Relationship with familial caregivers | Baseline and 6 months
  Change from baseline to 6 month assessment in relationship with familial caregivers assessed using the Perception of Parents Scale
Self-efficacy | Baseline and 6 months
  Change from baseline to 6 month assessment in confidence with regard to control of psychotic symptoms assessed using the Self-Efficacy Scale for Schizophrenia
Experience of Stigma | Baseline and 6 months
  Change from baseline to 6 month assessment in experience of stigma with regard to mental illness assessed using the Stigma Questionnaire
quality of life | Baseline and 6 months
  Change from baseline to 6 month assessment in quality of life assessed using the WHO Quality of Life Scale-Brief
stage of recovery | Baseline and 6 months
  Change from baseline to 6 month assessment in stage of recovery with regard to mental illness assessed using the Stages of Recovery Instrument
Coping skills | Baseline and 6 months
  Change from baseline to 6 month assessment in level of coping skills assessed using the Ways of Coping Questionnaire
Time perspective | Baseline and 6 months
  Change from baseline to 6 month assessment in time orientation assessed using the Zimbardo Time Perspective Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Breitborde, Ph.D., Principal Investigator — The Ohio State Univerity
Locations (1):
- University of Arizona Department of Psychiatry, Tucson, Arizona, United States